CLINICAL TRIAL: NCT03152916
Title: Application of 3D Printing Technology in Subtalar Arthrodesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Xiaojun Duan, Deputy Director of the Center for Joint Surgery, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CfJSSouthwestH
Record Dates: First submitted 2017-05-05; First posted 2017-05-15 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Ankle Injuries
Keywords: subtalar joint; arthrodesis; 3d printing
MeSH Terms: conditions — Ankle Injuries; Ankylosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D printing personalized plate (Experimental): 3D printing personalized plate will be used to guide the Kirschner wires in the joint fusion surgery.
  Interventions: Device: 3d printing personalized plate

INTERVENTIONS:
Device: 3d printing personalized plate — 3d printing personalized plate will be used in the subtalar arthrodensis

SUMMARY:
This study aims to use 3D printing personalized plate to locate the position in which the K-wires would be drilled to save operation time and decrease the number of times that the K-wires are drilled.

DETAILED DESCRIPTION:
Subtalar arthrodesis is a standard procedure for treating joint injuries in terminal stage. In this study, in order to improve efficacy and shorten the operation time, personalized plate is prepared before surgery. During the surgery, the articular cartilage is scraped, then the fusion joint is reset to the functional position; the 2-2mm Kirschner wires are drilled with the assistance of the personalized plate,then the position of the fusion joint as well as the Kirschner wires are confirmed under the C-arm; lastly, cannulated screws are screwed in along the Kirschner wires for effective fixation.

In the past surgeries without personalized plate, surgeons could only rely on their experience to locate the position for drilling and then confirm under the C-arm. This would prolong the operation time and be more traumatic to the patients. Using 3D printing personalized plate can solve this problem.

The preparation procedure for the personalized plate: firstly, ankle model are established according to the patient's CT scan data, then select modular pieces to prepare the personalized plate, sterilize it for future use. Apply conventional surgical treatment to the subtalar surface, reset the fusion joint to the functional position, and drill 2-2mm Kirschner wires with the guidance of the plate. If the locations of the fusion joint and the Kirschner wires are satisfying under the C-arm inspection, drill the hollow screw for final fixation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive subtalar arthrodesis and consider internal fixation with screws

Exclusion Criteria:

* Patients who receive subtalar arthrodesis but do not consider internal fixation with screws

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Operation time | Intraoperative
  Operation time for internal fixation

SECONDARY OUTCOMES:
Postoperative subtalar VAS score | Postoperative 1,6,12 months
  Postoperative subtalar VAS score of the patients
Fusion rate | Postoperative 1,6,12 months
  Fusion rate of the subtalar joint

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Duan, MD, Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang C, Cao J, Zhu H, Fan H, Yang L, Duan X. Endoscopic Treatment of Symptomatic Foot and Ankle Bone Cyst with 3D Printing Application. Biomed Res Int. 2020 Dec 26;2020:8323658. doi: 10.1155/2020/8323658. eCollection 2020. PMID 33426066